CLINICAL TRIAL: NCT00984321
Title: A Pilot Study of Geriatric Specific Interventions for Quality of Life in Elderly Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Joan Karnell Cancer Center at Pennsylvania (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-116
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Lymphoma Cancer; Gynecological Cancers
Keywords: Geriatric; Elderly; Counseling; Depression; Anxiety; Intervention; Psychoeducational; 09-116
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

ARMS (3):
- Psychoeducational Intervention Group (Experimental)
  Interventions: Behavioral: individual phone intervention and questionnaires
- Expressive Writing Intervention (Experimental)
  Interventions: Behavioral: expressive writing (arm will not be include in the randomization)
- Control Group (Active Comparator)
  Interventions: Behavioral: group intervention and questionnaires

INTERVENTIONS:
Behavioral: group intervention and questionnaires — Group Session will be 90 minutes long. Both the group sessions and individual session will be audio recorded. GSPI is a novel, manualized psychoeducational intervention that integrates Folkman's cognitive construct and Erikson's developmental concept of the 7th and 8th stages of life. GSPI consist of 5 weekly sessions. The first 2 sessions will be held on consecutive weeks to help establish rapport and explain therapeutic concepts, and next 3 sessions will be held every other week, giving patients time to utilize the therapeutic concepts and expanding length of contact with the patient.
  Arms: Control Group
Behavioral: individual phone intervention and questionnaires — Individual phone sessions will be 45 minutes long. Both the group sessions and individual session will be audio recorded. GSPI is a novel, manualized psychoeducational intervention that integrates Folkman's cognitive construct and Erikson's developmental concept of the 7th and 8th stages of life. GSPI consist of 5 weekly sessions. The first 2 sessions will be held on consecutive weeks to help establish rapport and explain therapeutic concepts, and next 3 sessions will be held every other week, giving patients time to utilize the therapeutic concepts and expanding length of contact with the patient.
  Arms: Psychoeducational Intervention Group
Behavioral: expressive writing (arm will not be include in the randomization) — intervention facilitate "reappraisal" through the exploration of past life events and prior successful ways of coping. Preliminary studies examining the efficacy of this writing intervention have shown its' ability to introduce patients to a new and effective coping method that can be utilized during future stressful cancer and aging related events.67 In the sessions, Wwe will explore past life events and ways of coping through manualized writing sessions.
  Arms: Expressive Writing Intervention

SUMMARY:
The purpose of this study is to examine whether psychoeducation counseling for older cancer patients undergoing treatment is feasible and worthwhile. The investigators will test this in a group or individual phone counseling format. Many cancer patients seek counseling to help with the emotional burden of their illnesses. Counseling often helps them cope with cancer by giving them a place to express their feelings. This geriatric-specific psychoeducation is intended to help older cancer patients cope with the burden of cancer and aging. The purpose of this study is to see if this type of counseling helps reduce depressive symptoms, anxiety, perception of loneliness and isolation. In addition this counseling aims to improve coping and quality of life (QOL).

Individuals who choose not to take part in the intervention study will be asked if they are willing to participate in a brief refusal sub study. The purpose of the refusal substudy is to compare levels of distress in patients that choose to participate and those that decline. This will yield valuable data that will help us distinguish between patients that decline due to lack of interest in research and those that decline due to high levels of distress. Participation in the refusal sub study consists of completion of 2 brief questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of prostate, breast cancer lung, lymphoma, or gynecological.
* Are receiving active treatment (e.g., radiation, hormone, or chemotherapy)or have been receiving treatment in the past 6 months for prostate, breast, lung, lymphoma, or gynecological cancer
* Are 70 years old or older
* Greater than 6-months post diagnosis
* Have a Distress Thermometer score of 4 or greater or

a score of ≥ 6 on the Depression or Anxiety subscale of the HADS

* Have a Karnofsky Performance Rating of 60 or greater
* In the investigator's judgment, participants must have satisfactory cognitive function to provide valid informed consent and participate in Geriatric Specific Psychoeducational Intervention. The Blessed Orientation-Memory-Concentration test (BOMC) will be used as a cognitive screening tool. Patients must have a BOMC score of less than or equal to 11.
* Able to converse, write and read in English. The questionnaires were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require a very lengthy process of reestablishing the reliability and validity and the establishment of norms for these measures. Therefore, participants must be able to communicate in English to complete the questionnaires.

Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in the intervention (e.g., acute psychiatric symptoms which requires individual treatment).
* As per self-report or review of the patient's medical record, if the patient is taking anti-depressant medication, fewer than three months on the same dose of anti-depressant medication.
* Actively participating in protocol 07-094 or 11-021

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
To test the feasibility, tolerability and acceptability of a Geriatric Specific Psychoeducational Intervention (GSPI) by examining the rates of eligibility, acceptance, and adherence. | 2 years

SECONDARY OUTCOMES:
To examine the impact of these GSPI in both formats on depressive symptoms, anxiety, demoralization, coping, loneliness and isolation, and spirituality compared to the control group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Joan Karnell Cancer Center at Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Tutino RC, Saracino RM, Kelman J, Schofield EA, Roth AJ, Nelson CJ. Cancer and aging: Reflections for elders- Expressive writing intervention: A pilot study. J Geriatr Oncol. 2022 Jun;13(5):706-714. doi: 10.1016/j.jgo.2022.02.009. Epub 2022 Mar 2. PMID 35246404
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm